CLINICAL TRIAL: NCT03088631
Title: Role of Metformin in Prevention of Premature Luteinization in Intracytoplasmic Sperm Injection Cycles
Brief Title: Metformin in Intracytoplasmic Sperm Injection Cycles
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reda S. Hussein, Lecturer of obstetrics and gynecology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MICSI
Record Dates: First submitted 2017-03-18; First posted 2017-03-23 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-04

CONDITIONS: Intracytoplasmatic Sperm Injection
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Eligible women who gave their informed consent were randomized into two groups: (I) metformin group and (II) placebo group. Randomization was conducted using a computer generated table of random numbers with allocation concealment. Randomization was not changed after it had been done.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Active Comparator)
  Interventions: Drug: Metformin
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — will receive metformin (1500 mg/day) starting with the commencement of oral contraceptive pills in the preceding cycle until the day of human chorionic gonadotropin triggering.
  Arms: Metformin group
Other: Placebo — will receive corn-flour placebo tablets (three tablets daily).
  Arms: Placebo group

SUMMARY:
The relationship between serum progesterone level on the day of human chorionic gonadotropin administration and outcome of in vitro fertilization /intracytoplasmic sperm injection and embryo transfer has been controversial for several decades. some studies presented data against the negative effect of premature luteinization and reported that elevated serum progesterone had no adverse effect on pregnancy rates in fresh embryo-transfer cycles within different ovarian responses. However, most studies have evaluated the association between serum progesterone level and clinical outcome in fresh in vitro fertilization /intracytoplasmic sperm injection cycles and advocated that serum progesterone elevation on the day of human chorionic gonadotropin administration may adversely affect the clinical outcome by jeopardizing endometrial receptivity.

In addition, the underlying mechanism through which premature luteinization influences clinical outcomes is elusive. some proposed that premature luteinization cause impairment of the endometrial receptivity, which may indicate a change in the implantation window, is more likely to be affected than the oocyte.whereas some documented that the compromised quality of oocytes might also be a cause.

The cut-off point of premature luteinization is not well established until now. Premature luteinization has been variously defined based on serum P levels, with thresholds of 0.9-1.5 ng/mL being used.

Previous studies have shown that metformin inhibits the first steps of steroidogenesis dose-dependently reducing granulosa cells progesterone output. Moreover, other authors have recently reported that low dose metformin could improve in vitro fertilization outcome in non poly-cystic ovarian syndrome repeaters. So, considering the safety of this drug before pregnancy, metformin can be given to consenting patients from first ultrasound monitoring until ovulation triggering.

ELIGIBILITY:
Inclusion Criteria:

* First or second trial ICSI cycle.
* Age: 20 -38 years
* BMI: patients with BMI ≥ 30 kg/m2 were advised to lose weight for 6 months through lifestyle modifications.
* AMH ≥1 ng/ml
* Basal FSH < 10 IU/ml.
* Normal uterine cavity evidenced by HSG or office hysteroscopy
* Normal levels of prolactin and TSH before starting COS cycle

Exclusion Criteria:

* Patients with recurrent two or more failed intra-cytoplasmic sperm injection cycles.
* Uterine anomalies or Synechiae.
* Severe male factor infertility
* Patients known to have diabetes, renal, liver disease, alcoholism, or drug abuse were excluded
* Patients who were on metformin treatment were asked to have a one month washout period before study participation.
* Poor responders

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of premature luteinization in both groups | 12 days
  Serum progesterone measurement ≥ 1.5 ng/ml by Mini-vidas assay was used to diagnose cases of premature luteinization.

SECONDARY OUTCOMES:
ongoing pregnancy rate | 12 weeks
  The number of cases with pregnancy more than 12 weeks of gestation divided by the cycles initiated per 100.
Good quality embryo rate | 20 days
  The number of good day 3 embryos per all two-pronuclear embryos.
Progesterone-to-mature oocyte index (PMOI) | 17 days
  calculated by dividing the serum P level (ng/ml) by the number of mature oocytes.
Progesterone/estradiol ratio | 12 days
  calculated as [progesterone (ng/mL) × 1000]/esatradiol (pg/mL)
Implantation rate | 7 weeks
  The number of gestational sacs observed by trans-vaginal ultrasound divided by the number of embryos transferred.

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hussein RS, Elnashar I, Amin AF, Zhao Y, Abdelmagied AM, Abbas AM, Abdelaleem AA, Farghaly TA, Abdalmageed OS, Youssef AA, Badran E, Abou-Taleb HA. Effect of Metformin on Premature Luteinization and Pregnancy Outcomes in Intracytoplasmic Sperm Injection-Fresh Embryo Transfer Cycles: A Randomized Double-Blind Controlled Trial. Int J Fertil Steril. 2021 Apr;15(2):108-114. doi: 10.22074/IJFS.2020.134643. Epub 2021 Mar 11. PMID 33687163